IRAS ID: 152483

<To be printed on hospital headed paper>

Study title: A Phase I/II, Dose Escalation Study to Assess the Safety and Tolerability of VAL201 in Patients with Locally Advanced or Metastatic Prostate Cancer and Other Advanced Solid Tumours

Dose finding safety study of VAL201 in cancer patients

#### PARTICIPANT INFORMATION SHEET AND CONSENT FORM

You are being invited to take part in a research study using an experimental (or investigational) drug called VAL201.

Before you decide whether to take part, it is important for you to understand why the study is being done and what it will involve.

Please take as much time as you need to read the following information carefully and discuss it with friends, relatives and your GP if you wish. Please ask us if there is anything that is not clear or if you would like more information. It is important that you take your time to decide whether or not you wish to take part.

There are 2 parts to this document:

- Part 1 This is to tell you about the study (why it is being done, how it will be carried out, possible benefits and potential risks of taking part) and what you will be expected to do. It will also explain how your medical information will be used and who may see it. If there is anything that is not clear or if you would like more information, you are free to ask us as many questions as you like.
- **Part 2** This provides more information on the study. If you agree to take part, you will be asked to sign an Informed Consent Form. You are free to change your mind and withdraw from the study at any time, without giving a reason.

A copy of this Participant Information Sheet and signed Informed Consent Form will be given to you to keep.

## Part 1

#### 1 Why is this study being done?

This study is the first in human study of the drug VAL201, which means it has never been given to humans before.

The main purpose of this study is to find the maximum dose that can be given to patients with either prostate cancer or other hormonally driven tumours. VAL201 is a manmade peptide (or small protein) which is intended to treat hormone-sensitive tumours by blocking the tumour cells normal hormone driven activity without affecting the patient's sexual hormone function. VAL201 is intended to interfere with the cells of the tumour, inhibiting them from their normal reproduction and the creation of new tumour cells. It is natural for cells to produce new cells whilst the older cells die. It is hoped that by slowing and stopping the creation of new cells, the size of the tumour will reduce.

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

Participants will be given weekly doses of VAL201 over a 21-day cycle. The study aims to assess patients over 6 cycles of treatment and any side effects will be closely monitored. The aim of the study is to gradually increase the dose over groups of patients. Each dose will need to be shown to be safe and well tolerated before the study moves onto the next dose level.

In addition to finding the maximum safe dose, the study will also investigate how VAL201 is absorbed, distributed, and removed from the body by evaluating the drug levels in the blood. There will also be assessments into how well VAL201 is able to prevent or slow the growth of the cancer tumour, and other biological effects on the body and the tumour.

### Why have I been invited?

You have been identified by your cancer consultant/oncologist as being suitable for this study. Eligible patients have locally advanced or metastatic prostate cancer or other advanced solid tumours. A locally advanced cancer is one that has started to spread to nearby tissues and a metastatic cancer has spread to other parts of the body.

Up to 42 male and female patients aged 16 years or over, will be invited to take part in this study.

## 3 Do I have to take part?

Your participation is entirely voluntary, which means it is up to you to decide whether to join the study. Once you are happy that you understand this Participant Information Sheet and if you agree to take part, you will be asked to sign an Informed Consent Form. You are free to change your mind and withdraw at any time, without giving a reason. This will not affect the standard of care you receive.

### 4 What will happen to me if I take part?

You will be invited for a screening visit to review the study and to assess your eligibility for the study. If you decide to take part in the study a study doctor or nurse (as appropriate) will talk you through the study and you will be asked to sign a study consent form. The screening assessments can take place up to 28 days before you receive your first dose of drug.

Once confirmed as eligible you will progress onto the study to receive doses of VAL201 once a week on a 21-day cycle. It is hoped that you will receive up to 6 cycles of treatment if your tumour is responding well to treatment. Your physician will inject VAL201 subcutaneously (or just under your skin) in up to 4 sites (depending on the dose) most likely your upper arm, thigh or stomach region. The intended drug doses on the study are expected to range from 0.5mg/kg (based on your weight) to a maximum of 16.0mg/kg.

The dosing will continue if your tumour is responding to treatment for 6 cycles (though treatment may carry on past 6 cycles if you are doing well and your doctor feels you may benefit). If your physician feels that you are not benefiting, your treatment will be stopped and you will be invited to return 30 days after the last dose of drug for a final assessment.

From the screening visit to the final assessment, the study could take up to 6 months. If the study drug results show that the growth of your tumour has slowed or halted and your study doctor feels you may benefit, you may be allowed to continue taking the study drug after this study completes.

At the time of publishing this document, the study drug has been safely administered to 12 patients. The most common side effects recorded are an injection site reaction and fatigue. You will be closely monitored by the study team and a number of assessments performed at each study visit. Please see the following table for a list of clinic visits and assessments to be conducted (Table 1 for screening to Cycle 6 and Table 2 for clinic visits for Cycle 7 onwards):

PIS and ICF version: 6.0 dated 05 August 2019 

Table 1 - Study Schedule and Assessments - Screening to Cycle 6

| | | CYCLE 1 | | | | C | YCLI | E 2 | CYCLE 3 | | | | CYCLE 4 | | | | CYCLE 5 | | | CYCLE 6 | | | | FINAL<br>CYCLE<br>VISIT | FINAL<br>VISIT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day | Day | | | | Day | | | Day | | | | Day | | | | Day | | | Day | | | | C6D22 | |
| | -28<br>to 0 | 1 | 2 | 8 | 15 | 1 | 8 | 15 | 1 | 2 | 8 | 15 | 1 | 2 | 8 | 15 | 1 | 8 | 15 | 1 | 2 | 8 | 15 | | |
| Informed consent | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Patient information and demographics (ethnic origin/race, sex etc.) | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Review of medical history (prior diseases and illnesses) | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Assessment of disease and how it affects patients daily life (ECOG) | X | | | | | X | | | X | | | | X | | | | X | | | X | | | | X | X |
| Physical examination (including height and weight) | X | X | | X | X | X | X | X | X | | X | X | X | | X | X | X | X | X | X | | X | X | X | X |
| Vital signs (heart rate/pulse, blood pressure, temperature and breathing rate) | X | X | | X | X | X | X | X | X | | X | X | X | | X | X | X | X | X | X | | X | X | X | X |

| Electrocardiogram – review of heart function | X | X | | | | X | | | X | | | | X | | | | X | | | X | | | | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Blood samples | X | | X | X | X | X | X | X | X | | X | X | X | | X | X | X | X | X | X | | X | X | X | X |
| Urine Collection & Pregnancy test (females only) | X | X | | | | X | | | X | | | | X | | | | X | | | X | | | | | |
| Tumour assessment (CT scan or MRI scan, and bone scan every three cycles) | X | | | | | | | | | | | | X | | | | | | | | | | | (X) | (X) |
| Tumour assessment (PSA blood test) | X | X | | | | X | | | X | | | | X | | | | X | | | X | | | | (X) | (X) |
| Tumour tissue sample/biopsy (optional) | (X) | | | | | | | | | | | | | | (X) | · | | | | | | <u>'</u> | | | |
| Review of side<br>effects and<br>ongoing subject<br>health | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Review of non-<br>study medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Dosing of study drug (VAL201) | | X | | X | X | X | X | X | X | | X | X | X | | X | X | X | X | X | X | | X | X | | |

IRAS ID: 152483

#### **Footnotes**

- Additional assessments may be conducted as clinically indicated.
- (X) denotes an assessment that is optional. The study team will be asking you separately whether you consent to this specific assessment
- Blood samples will be taken to check your health during screening and on Day 1 of each cycle and at the final study visit;
- Blood samples to investigate study drug levels may be taken at:
  - Cycle 1 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 6 Day 1: Pre-dose (0h) then 5, 10, 15, 30, 60, 90 min, 2, 3, 4, 5, 6, 8 h post-administration
- Blood samples for how study drug is affecting you and your tumour (up to 7 samples) will be taken in the study, at screening and Day 15 of every cycle of treatment up to Cycle 6.

As the study progresses, the Sponsor may decide to alter when the study dosing and assessments are to be performed compared to the above summary. In this case you will be provided with a separate table listing the visits and the assessments to be conducted.

Table 2 – Study Schedule and Assessments –Cycle 7 onwards

| | Cycl | Final | | |
|---|---|---|---|---|
| | | Day | | Study |
| | 1 | 8 | 15 | Visit |
| Assessment of disease and how it affects patients daily life (ECOG) | Х | | | Х |
| Physical examination | Х | | | Х |
| Vital signs (heart rate/pulse, blood pressure, temperature and breathing rate) | Х | | | Х |
| Electrocardiogram – review of heart function | Х | | | Х |
| Blood samples | Х | | | Х |
| Pregnancy test (females only) | Х | | | |
| Tumour assessment every 4 cycles (CT scan or MRI scan, and bone scan – disease specific) | Х | | | (X) |
| Review of side effects and ongoing subject health | Х | Х | Х | Х |
| Review of non-study medications | Х | Х | Х | Х |
| VAL201 administration | Х | Х | Х | |

#### **Footnotes**

Additional assessments may be conducted as clinically indicated.

#### *Review of Medical History and Non-study Medications*

At the start of the study you will be asked to provide information about your medical history and a list of medications including any current or past drugs, any herbal therapies, any self-medications such as multivitamins and minerals and any over the counter medications you may be taking for pain, cold or allergies. At all subsequent visits, if your condition and/or medications change during the course of the study, you will need to inform the study staff of these changes.

## Disease assessment and effect on daily life

The Eastern Cooperative Oncology Group (ECOG) performance scale is used by doctors and researchers to assess how a patient's disease is progressing. It will be used to assess how your disease affects your daily living abilities throughout the study.

#### **Physical Examination**

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

This will include an examination of your general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and tests on your nervous systems (e.g., eye movement, knee jerk). Height and weight will also be measured at screening with weight checks taken over the study.

## Vital Sign Assessment

Vital signs measurement (including your temperature, breathing rate, blood pressure, and heart rate/pulse) will be obtained.

## Electrocardiogram (ECG)

An electrocardiogram will be used to measure the electrical activity of your heart.

### **Blood Samples**

Blood samples will be taken over the course of the study and will include various tests to check your health and to check for the study drug levels in your blood. Additional blood samples will be taken to assess how VAL201 is affecting both you and the tumour. These samples will be destroyed after completion of the study.

All tests performed for safety measures such as standard haematology and blood chemistry will be analysed at a local laboratory. The samples will be handled and destroyed after analysis according to the local laboratory standard procedures.

Blood samples for all other analyses will be stored and sent outside of the hospital to specialized secure laboratories for analysis. The samples will be sent coded, thus your identity can only be traced back to you through the study site personnel who will keep a code list.

#### **Urine Collection**

Urine samples will be taken for various tests to check your ongoing health. These samples will be analysed locally at your hospital and will be handled and destroyed after analysis according to the local laboratory standard procedures.

#### Pregnancy testing

For female participants only, there will be regular pregnancy testing. The analysis will be conducted on blood or urine collected as part of your safety assessments.

#### <u>Tumour Assessment – disease assessments</u>

The status of your tumour will be checked by MRI scans or CT scans; if you are a prostate cancer patient you may also have radionuclide bone scans to assess the tumour.

- 1) Whole body radionuclide bone scan (Prostate cancer patients only)- A bone scan involves injecting a radioactive material (radiotracer) into a blood vein. The substance travels through your blood to the bones and organs. As it wears off, it gives off a little bit of radiation. This radiation is detected by a camera that slowly scans your body. The camera takes pictures of how much radiotracer collects in the bones and will be used to show any bone lesions or metastatic tumours in your bones.
- **2) CT scan (computerised tomography)** A CT scan uses X-rays and a computer to create detailed images of the inside of the body. You'll be exposed to radiation in the form of X-rays from your chest down to the tops of your legs (pelvis) to assess your tumour.
- *MRI (Magnetic resonance imaging)* An MRI scan uses a large magnet and radio waves to look at organs and structures inside your body to assess your tumour.
- *4) Prostate cancer patients only* Prostate-specific Antigen blood analysis will be conducted for patients with prostate cancer only to assess their disease status. This analysis

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

forms part of the blood sampling that is conducted locally at your hospital throughout the study.

# Optional Tissue Sampling - Biopsy collections

**New tumour tissue samples** - the provision of tumour tissue samples or biopsy samples is completely optional to you. If you decide not to consent to the procedures to obtain such samples, your involvement in the study or future medical care will not be affected. The tissue samples will be taken for the assessment of biological activity of the study drug in the tumour tissue. If you provide consent to have tissue samples collected, after you have received an anaesthetic (the area will be numbed or the lower part of your body will be numbed with an injection at your spine), your doctor will look at your tumour and snip small pieces (biopsies) of it for storage and testing later in the laboratory. Imaging may be used to help locate the tumour when collecting the tissue sample. Two samples will be collected, one prior to the start of study drug e.g. at screening and one after treatment has commenced in Cycle 3 Day 15. During the study, the tissue samples will be stored in a secure laboratory, with a sub-sample prepared for storage and future evaluation of study drug. After completion of the study analysis of these samples, if there is any remaining tissue it will be returned to your local hospital for your Doctor to use to support your future medical treatment.

If you do agree to provide a biopsy sample an additional 10 ml blood sample will be taken to enable a genetic comparison of your body's normal DNA to the tumour cell DNA. The results of the tests for this optional part are for research purposes only investigating mutations in tumour cell DNA. The results will not be of individual significance to you and they will not be used for your medical care. Therefore, results will not be provided to you or your study doctor.

Access to previously collected tumour tissues samples—if you have previously had a biopsy of your tumour we may ask you to consent to have access to part of this sample tissue for study testing. The study Sponsor will only request access to this historical tissue sample from your doctor following specific written approval from yourself to do so. After completion of the study analysis of this sample, if there is any remaining tissue it will be returned to your local hospital for your Doctor to use to support your future medical treatment.

If you do agree to provide a biopsy sample from tumour tissue that you have previously provided prior to this study, an additional 10 ml blood sample will be taken to enable a genetic comparison of your body's normal DNA to the tumour cell DNA. The results of the tests for this optional part are for research purposes only investigating mutations in tumour cell DNA. The results will not be of individual significance to you and they will not be used for your medical care. Therefore, results will not be provided to you or your study doctor.

#### Review of Side Effects and Ongoing Subject Health

Throughout the study you will be asked how you feel and will be encouraged to report to your study doctor if you feel unwell at any time. You will be given a card with contact details of your study doctor who you can contact to report any effects you are feeling throughout the study up until your final study assessment visit.

### Study Visits and Dosing Days

The diagram below summarises the expected number of visits and the study design. The starting dose of VAL201 was 0.5 mg/kg (0.5 mg per every kg you weigh) in the first cohort of patients, and as the study progresses to the  $6^{\text{th}}$  cohort of patients, the dose will not exceed 16.0 mg/kg. You will receive doses of VAL201 once a week on a 21-day cycle.

For Cycles 1, 3, 4 and 6 you will attend for visits on Days 1, 2, 8 and 15 and during Cycles 2 and 5 you will attend for visits on Days 1, 8, 15.

If your doctor feels you are doing well and you are benefiting from treatment, you may continue

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

to receive Cycles of treatment on Days 1, 8 and 15 after Cycle 6. A Follow-up visit will be completed 30 days after your last dose of treatment.

Diagram 1 Summary of visits and dosing days Cohorts 5&6



## 5 Expenses and payments

The study sponsor ValiRx is providing the study drug VAL201 free of charge and will cover all other study related costs or procedures not considered part of standard care for someone with your illness. Reasonable travel costs (by public transport or car, including parking) arising from attending study visits will be reimbursed in exchange for a receipt. You will not be paid for participating in this study.

Your study doctor and study clinic/hospital are being paid by the study sponsor to conduct this research.

Any data or specimens (for example, blood, urine, tissue samples) collected during this study and stored after study completion, may be used in research or in the development of future products. The sponsor does not intend to provide you with ownership or financial benefits that may result from this research or future commercial products.

#### 6 What will I have to do?

You will be asked to attend the research unit for the screening visit and every assessment and dosing day as detailed in the study schedule (Table 1 or a separate schedule as provided to you by your research team) up until a final study assessment. However you may withdraw at any time or the study doctor may decide it is in your best interests to be removed from the study.

It is important that, at all times during the study, you tell the study staff if you have taken any other medications than those given to you for the purpose of this study or agreed with your study doctor. This includes any over-the-counter medications, vitamins, herbal supplements or dietary supplements. If you have to see another doctor or are admitted into the hospital, please let them know that you are participating in this study and show them the patient card you will receive from your study doctor. Please notify the study staff as quickly as possible of these types of events.

### 7 What are the alternatives for diagnosis or treatment?

Discuss with your doctor what other specific treatment options you have and your doctor will discuss the alternative treatments.

#### 8 What are the possible disadvantages and risks of taking part?

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

Before participating in this study, you should consider if this will affect any personal insurance e.g. life insurance/assurance you have and seek advice if necessary.

### Surgery: Tissue sampling / Tumour Biopsy

The surgical risks are similar to biopsies that you have previously had. These include a risk of bleeding and infection. In addition, there are risks associated with the anaesthesia used which may include feeling sick/nausea, vomiting, or infection at the site of the needle injection.

### Administration of study drug

The study drug VAL201, will be injected under the skin (subcutaneously) into most likely your upper arm, leg (thigh) or stomach (approximately an inch away from your belly button). You may experience some discomfort in the injection area. Please report all discomfort experienced to your study doctor.

#### Other Risks:

## Blood Sampling

Drawing blood results in local discomfort and may also cause bruising. No more than 631.5 ml (just over a pint) of blood will be drawn over the 6-month period from screening to the Final Study visit. Placement of a cannula (small plastic tube placed directly into the blood vein) is a routine procedure that involves momentary discomfort at the time of insertion. Minor bruising may occur. In rare cases, phlebitis (irritation of the vein), extravasation (leaking of fluid outside the vein), and infection can also occur which resolves with or without antibiotic treatment.

### <u>Electrocardiogram</u>

Some people have a skin reaction to the sticky electrode patches that attach to the chest for the electrocardiogram. This skin irritation usually disappears when the patches are removed. Some males may have some chest hair shaved to ensure adequate contact between the electrodes and the skin.

### Whole body radionuclide bone scan

The scan involves one injection but, apart from that, it is painless. To have the scan, you first have a radioactive substance called a radionuclide injected into your bloodstream.

Before you have the injection, the nurse or radiographer will ask you about allergies or asthma as some people can be allergic to it. The injection may make you feel hot and flushed for a minute or two. The doctor will ask you to pass urine just before you return (or when you return) to get rid of any radionuclide in your bladder. Otherwise this could interfere with the scan. When you are ready for the scan, you will lie down on an X-ray couch and will need to keep still. Your body goes through the scanner. This makes some people feel claustrophobic, so let your doctor or nurse know if you feel nervous as they can help to reassure you. The scan takes about an hour. The radiation dose of each bone scan is equivalent to about 14 months of natural background radiation. The risk of all the bone scans causing a cancer is about 1 in 1100. The body gets rid of the radionuclide in the urine. This takes up to 24 hours. If you need to take any precautions in the meantime, the doctor or nurses will tell you beforehand.

#### CT scan or MRI

A CT scan uses X-rays and a computer to create detailed images of the inside of the body. You'll be exposed to radiation in the form of X-rays for a full body scan. The radiation dose of each CT is equivalent to about 8 years of natural background radiation. The risk of all the potential CT scans including the possible CT biopsy causing a cancer is about 1 in 143.

These risks (from the bone scans and the CT scans) should be considered in the context of 1 in 4

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

naturally occurring risk and are the risks to the average population and not someone with your clinical condition. Therefore it is reasonable to say that the risk from the radiation from this study can be considered small.

An MRI is a type of scan that uses strong magnetic fields and radio waves to produce detailed images of the inside of the body. An MRI scan is a painless and safe procedure. You may find it uncomfortable if you have claustrophobia and are nor suitable for people who have certain types of implants. Please talk to your doctor if you have any questions or concerns about these tests.

#### Allergic Reactions

Rare or unknown side effects could possibly occur, including life-threatening reactions. As with any drug, it is possible that you could experience an allergic reaction, such as itching, skin rash, facial swelling, and an acute or sudden drop in blood pressure. The latter may lead to shock with loss of consciousness and/or possible seizures, including the possibility of death. If any of the above symptoms of an allergic reaction occurs, seek medical attention immediately.

Please remember that as with any drug, there is a risk that a rare or previously unknown side effect will occur.

# 9 What are the side effects of any treatment when taking part?

Patients that have received VAL201 in clinical study to date, have experienced the following side effects considered related to the VAL201 study drug:

- Injection site reaction (rash/redness/pain/tenderness/itching/bruising)
- Fatigue
- Raised blood pressure (hypertension)

If you experience any side effects that you are concerned about you should contact your study doctor immediately.

## <add study doctor contact details here>

#### Harm to the unborn child:

You must avoid becoming pregnant or fathering a child while participating in this study. If you are a woman that can bear children (that is, not surgically sterile or has not gone through menopause), there may be a possibility that the study drug may harm an unborn child or nursing infant. For this reason, if you are pregnant, plan to become pregnant, or are breast-feeding, you CANNOT take part in this study. By signing the consent form, you confirm to the best of your knowledge that you are not pregnant now, you are not currently breast-feeding and you do not intend to become pregnant or start breast feeding during the study. If at any time during this study you think you might be pregnant, or later learn that you were pregnant during the study or wish to start breast feeding, you must contact the study doctor immediately for further instructions regarding your participation in this study and follow-up. If you become pregnant at any time during the study you will be immediately withdrawn from the study.

If you are a woman that can bear children, you must have a negative blood pregnancy test at screening before you can enter the study. In addition, if you are a woman that can bear children, or a man whose female partner can bear children, you and your partner must BOTH be on a form of contraception during the treatment period and for at least 1month after the last dose of the study drug.

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

If you are a male patient, you should use an effective method of contraception method upon enrolment, during the course of the study, and for 1month following the last study drug dosing. In the case of the woman who can bear children (whether study subject or partner of the study subject), you/she must already be using an effective method of contraception (e.g. barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine device (a device which is placed within the uterus)).

In the case of the man (whether study participant or partner of the study subject), an effective form of contraception must be used.

## 10 What are the possible benefits of taking part?

It is possible that you may benefit from the care given and that your tumour may respond to the study treatment. VAL201 has not been tested in humans previously which means that there is no evidence that your treatment will be successful. You should not enrol in this study with any expectation that you will personally benefit, but your participation may help to provide information that will be useful for future patients needing treatment for tumours like yours.

Research provides wider benefits to society / others with a similar condition and some indirect benefits might be foreseeable for participants themselves.

## What happens when the research study stops?

If the study drug results show that the growth of your tumour has slowed or halted and your study doctor feels you may benefit, you may be allowed to continue taking the study drug for more than 6 cycles as part of this protocol. You will be expected to continue to attend study visits as required by your doctor so that your progress can be monitored.

#### What if there is a problem?

Any complaint about the way you have been dealt with during the study or any possible harm you might suffer will be addressed. The detailed information on this is given in Part 2.

### Will my taking part in the study be kept confidential?

Yes, we will follow ethical and legal practice and all information about you will be handled in confidence. The details are included in Part 2.

This completes part 1.

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

#### Part 2.

#### 1 What if new information becomes available?

Sometimes during the course of the study new information becomes available concerning the investigational drug. If this happens, your study doctor will tell you about it and discuss with you whether you want to continue in the study. Also on receiving new information your study doctor might consider it to be in your best interests to withdraw you from the study. He/she will explain the reasons why it is best that you do not continue on study and will arrange for your ongoing medical care.

### What happens if I don't want to carry on with the study?

Your decision to take part in this study is entirely voluntary, and you can change your mind at a later stage.

Any decision to withdraw (or to decline this invitation to take part) in this study will not affect the care you receive from any relevant service (e.g. for patients, from the NHS).

Information and data collected up until the time of your withdrawal of consent may still be used. Any stored blood or tissue samples already collected will remain the property of the study Sponsor until they are destroyed (blood) or returned to your local hospital for your Doctor to use to support your future medical treatment (tissue).

## 3 What if there is a problem?

If you have a concern about any aspect of this study, you should ask to speak to the study team who will do their best to answer your questions, <Dr Name> at Tel. No. <tel number>. If you remain unhappy and wish to complain formally, you can do this <add complaint procedure here>.

The Sponsor does not expect you to suffer any health problems by taking part in this study. However, the Sponsor will compensate any patient who suffers injury, which is attributable to this study in accordance with the Clinical Trial Compensation Guidelines published by the Association of the British Pharmaceutical Industry (ABPI), a copy of which is available on request.

If you experience a research injury, emergency medical treatment will be provided. A research injury is any physical injury or illness caused by administration of the Sponsor study medicine or any study procedure that would not have occurred but for your inclusion in the study.

NHS trusts will compensate for medical negligence on their part.

## 4 Will my taking part in the study be kept confidential?

ValiRx Plc, is the sponsor for this study based in the United Kingdom. We will be using information from you and your medical records in order to undertake this study and will act as the data controller for this study. This means that we are responsible for looking after your information and using it properly. ValiRx Plc, will keep identifiable information about you for a minimum of 15 years after the study has finished.

Your rights to access, change or move your information are limited, as we need to manage your information in specific ways in order for the research to be reliable and accurate. If you withdraw from the study, we will keep the information about you that we have already obtained. To safeguard your rights, we will use the minimum personally-identifiable information possible.

You can find out more about how we use your information at https://www.valirx.com/about-us/privacy-and-gdpr/ or contact <a href="mailto:George.morris@valirx.com">George.morris@valirx.com</a>.

[NHS site] will collect information from you and your medical records for this research study in

PIS and ICF version: 6.0 dated 05 August 2019 

Protocol Number: VAL201-001

ValiRx Plc

IRAS ID: 152483

accordance with our instructions.

[NHS site] will keep your name, NHS number and contact details confidential and will not pass this information to ValiRxPlc. [NHS site] will use this information as needed, to contact you about the research study, and make sure that relevant information about the study is recorded for your care, and to oversee the quality of the study. Certain individuals from ValiRx Plc and regulatory organisations may look at your medical and research records to check the accuracy of the research study. ValiRx Plc will only receive information without any identifying information. The people who analyse the information will not be able to identify you and will not be able to find out your name, NHS number or contact details.

[NHS site] will keep identifiable information about you from this study for at least 15 years after the study has finished.

When you agree to take part in a research study, the information about your health and care may be provided to researchers running other research studies in this organisation and in other organisations. These organisations may be universities, NHS organisations or companies involved in health and care research in this country or abroad. Your information will only be used by organisations and researchers to conduct research in accordance with the UK Policy Framework for Health and Social Care Research.

Your information could be used for research in any aspect of health or care, and could be combined with information about you from other sources held by researchers, the NHS or government.

Where this information could identify you, the information will be held securely with strict arrangements about who can access the information. The information will only be used for the purpose of health and care research, or to contact you about future opportunities to participate in research. It will not be used to make decisions about future services available to you, such as insurance.

Where there is a risk that you can be identified your data will only be used in research that has been independently reviewed by an ethics committee.

Throughout this study your doctors, nurses, and other study personnel will record information about you in forms provided by us (known as "case report forms"). This personal information will include information about your health and your demographic details (such as your date of birth, your sex, and your ethnic origin/race).

All records and all other information about you entered into the case report forms will be identified by a unique study participant number, not your full name.

The Sponsor may use the information collected by us:

- By storing and analysing it electronically to find out what this study is telling us;
- by sharing it with regulatory authorities that approve new medicines, or with groups that check that research is done properly:
- by publishing the results of the study (this will not include any information that directly identifies you):
- By sharing it as part of research with other companies or universities for the purpose of further understanding or developing this drug. If the information is sent to another country, ValiRx will apply the same level of protection to your information, to the extent permitted by local law;
- By using it to plan new studies or other types of research or other medical purposes related to the development of the drug.

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

By consenting to this study you understand that all data derived from this study or from the specimens or samples obtained from you are the properties of the study Sponsor. In the event you withdraw your consent to participate in the study, you may be asked if you will allow the continued analysis of your samples and specimens, collected up to the time you withdrew your consent and the data to be used in analyses. Your permission will be recorded in writing. However, as provided under applicable data protection law you have the right of access to data relating to yourself and if needed, correct such data. You have certain rights, which may allow you to have access to data held about you, and to object or prevent certain processing of your information if it will cause you damage or distress. You understand that you may obtain access to such data through your study doctor.

Monitors, auditors, ethics committees and the regulatory authorities will be granted direct access to your original medical records for verification of clinical trial procedures and/or data, without violating your confidentiality, to the extent permitted by the applicable laws and regulations.

By signing the written informed consent form you authorise such access. For further details on your rights and how you can enforce them, you should contact the Information Commissioner (Wycliffe House, Water Lane, Wilmslow, and Cheshire, SK9 5AF).

## 5 Involvement of the General Practitioner/Family doctor (GP)

With your consent your family doctor (General Practitioner) will be told that you have decided to take part in this study.

## 6 What will happen to the samples I give?

Your samples will be stored and used for the tests described in this Participant Information Sheet. Any excess blood samples will be destroyed by the Sponsor when the analysis has been completed. Any remaining tissue samples will be returned to your local hospital for your Doctor to use to support your future medical treatment.

Blood samples will be taken over the course of the study and will include various tests to check your health and to check for the study drug levels in your blood. Additional blood samples will be taken to assess how VAL201 is affecting both you and the tumour. Specifically there will be assessment of biomarkers on both blood and tissue samples. A biomarker is a biological molecule found in blood, other body fluids or tissues that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition.

You will be requested to provide a specific consent for the optional testing on archived and/or fresh tumour tissue where a sample is available.

## 7 What will happen to the results of the research study?

The study results will be published on a publically accessible database e.g. clinincialtrials.gov and may also be published in scientific journals, however in all cases, personal information identifying you as a participant will not be released.

#### 8 Who is organising and funding the research?

The study is sponsored by ValiRx plc. UK, a pharmaceutical company. This means that ValiRx plc is paying the research team for the costs of the study.

# 9 Who has reviewed the study?

PIS and ICF version: 6.0 dated 05 August 2019 

IRAS ID: 152483

The study protocol and this information sheet has been submitted to the UK Regulatory Authority (MHRA) and a registered Research Ethics Committee and these committees have approved this study. This study will be conducted under Good Clinical Practice guidelines (an international ethical and scientific quality standard for clinical trials involving human participants).

#### Further information and contact details

If you have any questions about this study, please contact your study doctor or other study personnel.

Contact details [add the details of Principal Investigator; if the PI is not the point of contact for the patient, modify accordingly]:

<Add study nurse's name and telephone number>

For any concerns about your rights as a participant or any complaints please contact:

<Add hospital/trust complaints department/patient services>

## For emergencies only please contact:

<Add 24hr emergency telephone number>

Before you sign the informed consent form, you should ask questions about anything that you do not understand. The study staff will answer any questions before, during and after the study.

Thank you for taking the time to read this information sheet.

PIS and ICF version: 6.0 dated 05 August 2019 

| | ValiRx Plc | Protocol Number: VAL201-0 | 001 |
|---|---|---|---|
| | IRAS ID: 152483 | | |
| | Centre Number: | | |
| | Study Number: VAL201-001 | | |
| | Patient Identification Number for this trial: | | |
| - | CONSENT FORM | | |
| V | itle of Project: A Phase I/II, Dose Escalation Study to Asse<br>AL201 in Patients with Locally Advanced or Metastatic P<br>dvanced Solid Tumours | | ility of |
| | Name of Researcher: [NAME OF INVESTIGATOR] | Plea | ise initial |
| | all boxes | | |
| 1. | I confirm that I have read and understand the information so (version [VERSION NUMBER]) for the above study. I have consider the information, ask questions and have had these | had the opportunity to | |
| 2. | I have been informed that there has been a change in the pl assessment schedule and have been provided with the new <b>NUMBER</b> ]) for reference. | • | |
| 3. | I understand that my participation is voluntary and that I a | m free to withdraw at any | |
| | time without giving any reason, without my medical care or | r legal rights being affected. | |
| 4. | I confirm to the best of my knowledge that I am not pregnant breast-feeding and do not intend to become pregnant or stated study. Not a | - | |
| 5. | I understand that relevant sections of my medical notes and study, may be looked at by individuals from ValiRx, from Vafrom regulatory authorities or from the NHS Trust, where it part in this research. I give permission for these individuals records. | aliRx authorised persons,<br>t is relevant to my taking | |
| 6. | I agree to take part in the above study. I agree that samples personal data, in anonymised form may be transferred and PIS for the study. | - | |

PIS and ICF version: 6.0 dated 05 August 2019

7. I agree to my GP being informed of my participation in the study.

IRAS ID: 152483

taking consent

Optional testing for tumour biopsy analysis - by initialing either of the following two boxes below I am specifically providing consent for the optional tumour analysis listed. If I decide not to consent to this testing, I understand that my involvement in the study or future medical care will not be affected.